CLINICAL TRIAL: NCT04254146
Title: Effects of Acute Exercise on BDNF Levels in Rheumatoid Arthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Research Assistant, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-04
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Brain Derived Neurotrophic Factor; acute exercise
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Aerobic exercise will be performed for a single session
  Interventions: Other: Aerobic exercise
- Control group (Active Comparator): Aerobic exercise will be performed to healthy population for a single session
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise will be performed to all participants for a single session. Maximum heart rate was calculated for each subject (220 - age) and a heart rate monitor (Polar FT 100, China) will be used to follow subjects' heart rate during aerobic exercise.

SUMMARY:
Background: RA may progress with articular and non-articular involvement.Depression prevelance is found to increase for RA patients according to healthy population and to be correlated with pain, decreased quality of life, fatigue and physical disability.BDNF level was found significantly lower in RA patients with depression. Aim of this study is to investigate the variation of BDNF levels following acute exercise and potential correlation between BDNF levels and depression.

Methods: This study included 30 RA patients and 30 age and sex matched healthy controls.Depression levels were evaluated with Beck Depression Inventory (BDI) and Hospital Anxiety and Depression Scale (HADS). Blood samples from all subjects were taken and centrifuged before and immediately after the exercise intervention.

DETAILED DESCRIPTION:
Background: Rheumatoid Arthritis (RA) is a chronic, inflammatory, rheumatic disease that genetic and environmental factors play role in its pathogenesis. There may be other symptoms caused by both the inflammation and the chronic disease effect, as well as the symptoms associated with the disease, such as depression, fatigue, physical inactivity and decreased quality of life. Major depression risk was revealed 16.8% of RA patients in a meta-analysis. Depression prevalence was found 38.8% by the assessment with Patient Health Questionnaire (PHQ-9) and between 14.8% and 48% by the assessment with Hospital Anxiety and Depression Scale. BDNF is a neurotrofic factor that may show healing, survival-promoting and protective effects on neurons in central and peripheral nervous system. Acute or chronic exercise programmes were found to increase BDNF levels in human and animal studies. Aim of this study is to investigate the variation of BDNF levels following acute exercise and potential correlation between BDNF levels and depression.

Methods: This study included 30 RA patients and 30 age and sex matched healthy controls.Patients who were aged between 18-65 years, got diagnosed according to American College of Rheumatology criteria and were being followed at Firat University Department of Rheumatology were included in the study. Also, patients who had regular exercise habits, malignancy, pregnancy, incorporation, took anti-TNF treatment, had changes of medical treatment in last 3 months, diagnosed with Fibromyalgia Syndrome and Osteoarthritis for lower extremity, had cardiac symptoms according to New York Heart Association and had dysfunction that can prevent physical activity were excluded from the study. Healthy participants who were aged 18- 65 years old and not to have exercise habits were included in this study. Participants included in the study were asked and recorded age, body mass index (BMI), smoking/ alcohol habits, duration of the disease, vocation and having another chronic disease. Next, depression levels were evaluated with Beck Depression Inventory (BDI) and Hospital Anxiety and Depression Scale (HADS). Blood samples from all subjects were taken and centrifuged before and immediately after the exercise intervention.Aerobic exercise was performed to all participants for a single session. Maximum heart rate was calculated for each subject (220 - age) and a heart rate monitor (Polar FT 100, China) was used to follow subjects' heart rate during aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged between 18-65 years,
* Patients who got diagnosed according to American College of Rheumatology criteria
* Patients who were being followed at Firat University Department of Rheumatology

Exclusion Criteria:

* Patients who had regular exercise habits, malignancy, pregnancy, incorporation,
* Patients who took anti-TNF treatment
* Patients who had changes of medical treatment in last 3 months
* Patients who diagnosed with Fibromyalgia Syndrome and Osteoarthritis for lower extremity
* Patients who had cardiac symptoms according to New York Heart Association
* Patients who had dysfunction that can prevent physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-10-02 (Estimated); Study Completion 2020-12-02 (Estimated)

PRIMARY OUTCOMES:
BDNF levels | 1 minute
  Blood samples from all subjects will be taken and centrifuged before and immediately after the exercise intervention. Obtained serums will be stored at the laboratories of Firat University.

SECONDARY OUTCOMES:
Beck Depression Inventory | 2 minutes
  Turkish version of Beck Depression Inventory (BDI) will be used to determine the depression levels of subjects. It consists of 21 items regarding pessimism, guilt, sleep, appetite and fatigue and each item is scored between 0 and 3. Higher scores shows the severity of depression.Score > 18 of BDI was considered as a cut-off value for depression.
Hospital Anxiety and Depression Scale | 2 minutes
  Hospital Anxiety and Depression Scale (HADS), developed by Zigmond and Snaith, determines anxiety disorders and depression among patients in nonpsychiatric clinics. It consists of 14 items and each item is scored from 0 to 3. Seven items are associated with anxiety and seven relate to depression. Score ranges from 0 to 21. Bjelland et al. identified score of 8 as a cut-off point.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman S Koca, Study Director — Firat University
Locations (4):
- Turkey (Türkiye) (4):
  - Gülnihal Deniz, Elâzığ
  - Songul Baglan Yentur, Elâzığ
  - Süleyman Serdar Koca, Elâzığ
  - Zübeyde Ercan, Elâzığ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimsholm O, Rantapaa-Dahlqvist S, Dalen T, Forsgren S. BDNF in RA: downregulated in plasma following anti-TNF treatment but no correlation with inflammatory parameters. Clin Rheumatol. 2008 Oct;27(10):1289-97. doi: 10.1007/s10067-008-0910-4. Epub 2008 May 17. PMID 18484150
- [Background] Szuhany KL, Bugatti M, Otto MW. A meta-analytic review of the effects of exercise on brain-derived neurotrophic factor. J Psychiatr Res. 2015 Jan;60:56-64. doi: 10.1016/j.jpsychires.2014.10.003. Epub 2014 Oct 12. PMID 25455510